CLINICAL TRIAL: NCT03233347
Title: A Phase II Trial of PET-Directed Therapy Using AVD (Doxorubicin, Vinblastine, and Dacarbazine) Plus Brentuximab Vedotin Induction Chemotherapy, With or Without Brentuximab Vedotin Plus Nivolumab, Followed by Nivolumab Consolidation for Patients With Previously Untreated Non-Bulky Limited Stage Hodgkin Lymphoma
Brief Title: Doxorubicin, Vinblastine, Dacarbazine, Brentuximab Vedotin, and Nivolumab in Treating Patients With Stage I-II Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-LY-1601; NCI-2017-01308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-LY-1601 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Ann Arbor Stage I Hodgkin Lymphoma; Ann Arbor Stage IA Hodgkin Lymphoma; Ann Arbor Stage IB Hodgkin Lymphoma; Ann Arbor Stage II Hodgkin Lymphoma; Ann Arbor Stage IIA Hodgkin Lymphoma; Ann Arbor Stage IIB Hodgkin Lymphoma; Classic Hodgkin Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin; Dacarbazine; Doxorubicin; Nivolumab; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (combination chemotherapy, nivolumab) (Experimental): Patients receive doxorubicin IV over 3-5 minutes, vinblastine IV over 3-5 minutes, and dacarbazine IV over >= 30 minutes, and brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients with PET-positive then receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. PET-positive patients then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. PET-negative patients receive nivolumab IV over 30 minutes on day 1 starting after AVD and BV treatment. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Dacarbazine; Drug: Doxorubicin; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Drug: Vinblastine

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; VLB

SUMMARY:
This phase II trial evaluates how well AVD (doxorubicin, vinblastine, dacarbazine) in combination with brentuximab vedotin and nivolumab work in treating patients with stage I-II Hodgkin lymphoma. Drugs used in the chemotherapy, such as doxorubicin, vinblastine, dacarbazine, and brentuximab vedotin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, and/or by stopping them from spreading. Targeted agent, such as nivolumab, may interfere with the ability of cancer cells to grow and spread by enhancing the immune system. Giving doxorubicin, vinblastine, dacarbazine, brentuximab vedotin, and nivolumab may improve survival of patients with stage I-II Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate progression-free survival (PFS) at 3 years in patients with previously untreated stage I or II non-bulky Hodgkin lymphoma (HL) who received doxorubicin, vinblastine, dacarbazine (AVD) plus brentuximab vedotin (BV) induction therapy followed by nivolumab (N)VB consolidation therapy.

SECONDARY OBJECTIVES:

I. To estimate the overall survival (OS) rate at 3 years in patients with previously untreated stage I or II non-bulky HL who received AVD plus BV induction therapy followed by NVB consolidation therapy.

II. To estimate the percentage of patients with untreated stage I or II non-bulky HL who are positron emission tomography (PET) positive versus PET negative after 3 cycles of AVD plus BV induction therapy.

III. To estimate PFS and OS at 3 and 5 years separately for patients who are PET negative versus PET positive after 3 cycles of AVD plus BV induction followed by NVB consolidation therapy.

IV. To estimate time to progression (TTP) in patients with previously untreated stage I or II non-bulky HL who received AVD plus BV induction therapy followed by NVB consolidation therapy.

V. To estimate the overall response rate and the number of patients who convert to complete response (CMR) after NVB in patients with partial response (PMR) at the end of AVD plus BV induction therapy.

VI. To estimate the duration of response in patients with previously untreated stage I or II non-bulky Hodgkin's lymphoma who received AVD plus BV induction therapy followed by NVB consolidation therapy.

VII. To evaluate the toxicity and tolerability of AVD plus BV induction followed by NVB consolidation therapy as assessed via the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version [v]4).

EXPLORATORY OBJECTIVES:

I. Optional biopsy tissue samples will be collected for future analysis. II. Optional blood sample will be collected for future analysis. III. Cost-benefit analysis of AVD plus BV followed by NVB consolidation, compared to the current standard therapy with adriamycin, bleomycin, vinblastine plus dacarbazine (ABVD) with or without radiation therapy.

OUTLINE:

Patients receive doxorubicin intravenously (IV) over 3-5 minutes, vinblastine IV over 3-5 minutes, and dacarbazine IV over >= 30 minutes, and brentuximab vedotin IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients with PET-positive then receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. PET-positive patients then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. PET-negative patients receive nivolumab IV over 30 minutes on day 1 starting after AVD and BV treatment. Treatment repeats every 2 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 and 8 weeks, every 3 or 6 months for 2 years, and then once a year for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease (>= 1.5 cm) as assessed by 2 dimensional measurement by computed tomography (CT)
* Previously untreated stage I or II non-bulky (defined as a mass measuring < 10 cm in the longest dimension by CT) classical Hodgkin lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Life expectancy >= 3 months
* Documented negative serologic testing for human immunodeficiency virus (HIV), hepatitis B (unless serologically positive due to prior vaccination), and hepatitis C =< 1 year prior to registration
* White blood cell >= 2,000 /mm^3 without transfusion support > 7 days prior to registration
* Hemoglobin >= 8.5 g/dL without transfusion support > 7 days prior to registration
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3 without transfusion support > 7 days prior to registration
* Platelet count >= 75,000/mm^3 without transfusion support > 7 days prior to registration
* Alanine and aspartate aminotransferase (ALT/AST) =< 2.5 x upper limit of normal (ULN) obtained =< 14 days prior to registration
* Total serum bilirubin =< 1.5 x ULN (if documented Gilberts syndrome =< 3 x ULN) obtained =< 14 days prior to registration
* Serum creatinine =< 1.5 x ULN or measured calculated creatinine clearance >= 40 ml/min for subject with creatinine levels > 1.5 x institutional ULN (per Cockcroft-Gault formula) obtained =< 14 days prior to registration
* Negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 7 days prior to registration in women of child-bearing potential (WOCBP)
* Sexually active female of reproductive capability ie, WOCBP, has agreed to use a medically accepted form of contraception from time of registration to completion of study therapy through 24 weeks (6 months) after last dose of NVB or BV; Note: Females of non-child-bearing potential are those who are postmenopausal for > 1 year or who have had a bilateral tubal ligation or hysterectomy
* Male subjects agree to use an adequate method of contraception starting with the first dose of study therapy through 31 weeks after the last dose of study therapy
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: During the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Prior therapies including involved field radiation therapy
* Bulky disease (defined as a nodal mass measuring >= 10 cm by CT)
* Known central nervous system (CNS) involvement
* Moderate or severe hepatic insufficiency Child-Pugh score > 6
* Severe renal impairment (i.e. creatinine clearance < 40 mL/min)
* Symptomatic cardiac disease including ventricular dysfunction, left ventricular ejection fraction < 45%, symptomatic coronary artery disease or symptomatic arrhythmias
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy =< 7 days prior to registration
* Known history of active TB (Bacillus tuberculosis)
* Requires therapy with agents that have a predisposition for hepatoxicity
* Hypersensitivity to NVB or any of its excipients or to any component of AVD + BV therapy
* Requires immunosuppressive doses of corticosteroid therapy (> 10 mg/day prednisone equivalents) for >= 2 weeks prior to registration
* Active, known, or suspected autoimmune disease that requires systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); Note: Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Active infection requiring systemic IV antibiotic therapy
* History of Steven's Johnson's syndrome, toxic epidermal necrolysis syndrome (TENs) or motor neuropathy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Received a live vaccine =< 30 days prior to registration; Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed; routine vaccinations, including seasonal influenza, must be given >= 2 weeks prior to registration
* History of allergies and adverse drug reaction to study drug components
* History of another primary malignancy that has not been in remission for at least 3 years; (Note: The following are exempt for the 3-year limit: nonmelanoma skin cancer, fully excised melanoma in situ [stage 0], curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on papanicolaou [PAP] smear)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of progressive promyelocytic leukemia (PML), known history of pancreatitis, active grade 3 or higher viral, bacterial or fungal infection =< 2 weeks prior to registration and documented history of cerebrovascular event (stroke or transient ischemic attack [TIA]) =< 6 months prior to registration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From registration, where progression is by computed tomography (CT)-based or positron emission tomography (PET)-CT based criteria, assessed at 3 years
  The distribution of progression-free survival time will be estimated using the method of Kaplan-Meier and the efficacy will be determined by the log rank statistic. Overall progression-free survival at 3 years will be reported.

SECONDARY OUTCOMES:
Overall survival | Time from registration to death due to any cause, assessed at 3 and 5 years
  The distribution of overall survival time will be estimated using the method of Kaplan-Meier. Will be estimated in each group.
The proportion of patients who are positron emission tomography (PET) negative | After 3 courses (84 days)
  Will be estimated by the number of patients who are PET negative divided by the total number of evaluable patients.
Proportion of patients who are positron emission tomography (PET) positive | After 3 courses (84 days)
  Will be estimated by the number of patients who are PET positive divided by the total number of evaluable patients.
Progression free survival | From registration, where progression is by CT-based or PET-CT based criteria, assessed at 84 days
  Differences between the groups will be assessed by log-rank statistics.
Progression free survival | From registration, where progression is by CT-based or PET-CT based criteria, assessed at 3 years
  Differences between the groups will be assessed by log-rank statistics.
Progression free survival | From registration, where progression is by CT-based or PET-CT based criteria, assessed at 5 years
  Differences between the groups will be assessed by log-rank statistics.
Overall response rate (ORR) | Up to 5 years
  The ORR will be estimated by the number of patients with an complete response (CR)/complete metabolic response/partial response (PR)/partial metabolic response or better divided by the total number of evaluable patients. The ORR may be analysed when all patients are off treatment. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Time to progression | Time from registration to the earliest date of documentation of disease progression, assessed up to 5 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
The proportion of patients who convert from partial response at the end of induction therapy to complete response after brentuximab vedotin plus nivolumab (NVB) | Up to 5 years
  Will be estimated by the number of patients who convert divided by the total number of evaluable patients who receive at least one dose of NVB induction therapy. Exact binomial 95% confidence intervals for the true conversion rate will be calculated.
Duration of response | Up to 5 years
  Will be defined for all evaluable patients who have achieved a PR or CR as the date at which the patient's objective status is first noted to be a response to the earliest date progression is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 5 years
  Will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Steven I Park, Principal Investigator — Academic and Community Cancer Research United
Locations (9):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center - Montlake, Seattle, Washington